CLINICAL TRIAL: NCT07383597
Title: A Randomized Pilot Study of LPS Adsorption Using the Efferon LPS Device in Patients With Ulcerative Colitis and Crohn's Disease During Disease Exacerbation
Brief Title: Lipopolysaccharide Adsorption (Efferon LPS) in Patients With Ulcerative Colitis and Crohn Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-lps-2025-04
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: Hemoadsorption; Hemoperfusion; Extracorporeal therapy; LPS adsorption
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Allocation of patients into groups will be done by stratified 1:1 randomisation.
  Each group will include an equal number of patients with Crohn's disease (n=10) and ulcerative colitis (n=10).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline therapy (No Intervention): These patients will receive standard therapy for Crohn disease or ulcerative colitis
- Baseline therapy + Efferon LPS (Experimental): These patients will receive standard therapy for Crohn disease or ulcerative colitis and Efferon LPS hemoadsorption.
  Interventions: Device: Efferon LPS

INTERVENTIONS:
Device: Efferon LPS — Efferon LPS, a medical device, which is a single-use cartridge filled with a polymeric adsorbent that selectively adsorbs endotoxin via surface-immobilized ligand and excessive cytokines via its intrinsic porosity.
  Hemoadsorption was administered in 3-4 sessions of at least 2 hours each via peripheral vascular access, with intervals of no more than 5 days between sessions.
  Arms: Baseline therapy + Efferon LPS

SUMMARY:
The goal of the study is to evaluate the safety and efficacy of multimodal (cytokine and lipopolysaccharide) hemoperfusion using the Efferon® LPS device in patients with ulcerative colitis and Crohn disease.

Participants will be assigned to two groups for comparison: a control group receiving baseline therapy and a treatment group receiving baseline therapy in combination with Efferon® LPS hemoadsorption.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) represent a group of chronic inflammatory disorders, with the main clinical entities being Crohn's disease and ulcerative colitis. The prevalence of IBD is increasing worldwide, imposing a substantial socioeconomic burden on society and healthcare systems.In IBD, in the presence of predisposing genetic factors and unclear triggers, a loss of immunological tolerance to luminal antigens occurs. This results in persistent inflammation of the intestinal wall, leading to mucosal damage and increased permeability of the mucosa to various antigens, which further amplify and sustain the pro-inflammatory immune response. Increased intestinal permeability and subsequent endotoxin translocation may also play a role in the pathogenesis of IBD.

Currently used treatments for IBD aim to control inflammation and modulate mucosal immune responses by blocking cytokine activity, such as tumor necrosis factor (TNF) and Interleukin 23, preventing the homing of immune cells to the gut, or inhibiting T-cell egress from lymph nodes.Steroid-free remission, due to the adverse effects associated with corticosteroids, is one of the primary treatment goals in IBD, whereas long-term corticosteroid use is considered a marker of suboptimal disease control.

Some patients with highly active IBD, who cannot be treated with pharmacological therapy for various reasons (including refractoriness, intolerance, or significant adverse effects), require alternative treatment approaches. Among these, extracorporeal therapy modalities, which have been rapidly developing in recent years, represent a promising therapeutic option.

Compared with standard steroid therapy, extracorporeal treatment modalities demonstrate comparable therapeutic efficacy and safety. In addition, extracorporeal therapies may represent an alternative treatment option for IBD without the undesirable adverse effects associated with systemic corticosteroids, immunosuppressants, and biologic agents. This also applies to hemoadsorption, which has been shown to reduce circulating levels of cytokines, various cytotoxins, myoglobin, and products of cellular breakdown in patients' blood. However, data on the use of cytokine hemoadsorption in IBD are extremely limited, and no published studies have been identified regarding the use of lipopolysaccharide (endotoxin) adsorption in IBD.

The Efferon® LPS device was originally developed for use in sepsis, leveraging its ability to effectively target both primary and secondary inflammatory mediators. This therapeutic approach also holds substantial potential for the treatment of other pathological conditions characterized by complex inflammatory responses.

This study aims to evaluate the safety and efficacy of multimodal (cytokine and lipopolysaccharide) hemoperfusion using the Efferon® LPS device in patients with ulcerative colitis and Crohn Disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease (ICD-10: K50), extensive disease, with a chronic continuous or relapsing course during an exacerbation (flare), including:

  * Severe flare: CDAI ≥ 450 and/or SES-CD > 15;
  * Moderate flare: CDAI 350-450 and/or SES-CD > 7, steroid-refractory.
* Ulcerative colitis (ICD-10: K51), with a chronic continuous or relapsing course during an exacerbation (flare), including:

  * Severe flare: Mayo score ≥ 10 and partial Mayo score ≥ 6;
  * Moderate flare: Mayo score 6-9 and partial Mayo score ≥ 3, steroid-refractory or steroid-dependent.
* Presence of signs and symptoms of ulcerative colitis or Crohn's disease for at least 3 months prior to study enrollment.
* The diagnosis must be confirmed by clinical and endoscopic findings and supported by a histopathology report
* The patient's condition allows Efferon LPS therapy to be performed for at least 2 hours

Exclusion Criteria:

* Indeterminate colitis, radiation colitis, ischemic colitis,confirmed presence of megacolon, strictures, or stenosis causing symptoms of intestinal obstruction.
* Expected need for bowel resection within 4 weeks after enrollment
* Presence at hospitalization of a stoma, ileal pouch-anal anastomosis, or a fistula with purulent discharge (which, in the investigator's opinion, is likely to require surgical or medical intervention within 4 weeks after enrollment), or planned ileostomy or colostomy.
* Partial or total colectomy, small bowel resection, or creation of a stoma (i.e., temporary or permanent colostomy, ileostomy, or other enterostomy) within 6 months prior to enrollment, or presence of an external or entero-enteric fistula with symptoms within 6 months prior to enrollment.
* Suspected or diagnosed intra-abdominal or perianal abscess that has not been adequately treated.
* Positive test for Clostridioides difficile toxin.
* Positive test for infectious pathogens (including helminth eggs, parasites, or bacterial infections).
* History of malignancy within the past 5 years, including solid tumors or hematologic malignancies (except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin in situ, or cervical dysplasia/cancer that has been surgically excised with complete resolution), or colonic mucosal dysplasia that has not been completely removed.
* End-stage renal disease.
* Acute pulmonary embolism confirmed by imaging.
* Acute myocardial infarction within the last 4 weeks.
* Acute cerebrovascular accident (stroke) within the last 8 weeks.
* Dementia.
* Uncontrolled bleeding (acute blood loss within the last 24 hours).
* History or current evidence of recurrent or chronic viral infection (e.g., hepatitis B virus, hepatitis C virus, or human immunodeficiency virus [HIV]).
* Alcohol or drug dependence.
* Any other condition that, in the investigator's opinion, would preclude the patient's participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Crohn's Disease Activity Index (CDAI) score | 1-90 days
  The Crohn's Disease Activity Index (CDAI) is calculated as a composite score based on a set of clinical and laboratory parameters reflecting disease activity. The higher the CDAI score, the greater the clinical activity of Crohn's disease. A CDAI score below 150 corresponds to clinical remission, scores of 150-300 indicate mild disease activity, 301-450 indicate moderate disease activity and a score of 450 points or higher is considered indicative of a severe disease flare.
Change in the Mayo score in patients with ulcerative colitis | 1-90 days
  The Mayo score is a composite index used to assess disease activity in ulcerative colitis. It includes four components evaluating stool frequency, rectal bleeding, endoscopic findings, and the physician's global assessment. Higher Mayo scores indicate greater severity of ulcerative colitis. Disease activity can be categorized based on the total Mayo score as follows: 0-2 points indicate remission, 3-5 points indicate mild disease, 6-9 points indicate moderate disease, and 10-12 points indicate severe disease.

SECONDARY OUTCOMES:
Change in the Simple Endoscopic Score for Crohn's Disease (SES-CD) | 1-90 days
  The Simple Endoscopic Score for Crohn's Disease (SES-CD) is an endoscopic index reflecting Crohn disease activity.The score is calculated as the sum of multiple endoscopic parameters assessed across different intestinal segments. Disease activity is classified as follows: 0-2 points - mucosal healing; 3-6 points - minimal activity; 7-15 points - moderate activity; ≥16 points - severe activity.
Change in the Endoscopic Activity Index for Ulcerative Colitis (Schroeder Score) | 1-90 days
  The endoscopic activity index for ulcerative colitis according to Schroeder (endoscopic Mayo subscore) is used to assess the severity of mucosal inflammation based on colonoscopic findings. The score ranges from 0 to 3 points, with higher values indicating greater endoscopic disease activity. A score of 0 corresponds to normal or inactive disease, a score of 1 indicates mild inflammatory changes, a score of 2 reflects moderate inflammation, and a score of 3 is characteristic of severe endoscopic activity with pronounced mucosal damage.
Hospital length of stay | 1-90 days
  Time (days) from enrollment to hospital discharge
The Inflammatory Bowel Disease Questionnaire (IBDQ) index | 1-90 days
  The Inflammatory Bowel Disease Questionnaire (IBDQ) is a validated disease-specific instrument used to assess health-related quality of life in patients with inflammatory bowel disease. It consists of 32 items grouped into four domains: bowel symptoms, systemic symptoms, emotional function, and social function. Each item is scored on a 7-point Likert scale, resulting in a total score ranging from 32 to 224 points, with higher scores indicating better quality of life. Changes in the IBDQ score over time reflect improvements or deterioration in patient-reported outcomes and overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Bakulin, PhD, MD, Principal Investigator — North-Western State Medical University named after I.I.Mechnikov
Locations (1):
- North-Western State Medical University named after I.I. Mechnikov, Saint Petersburg, Russia